CLINICAL TRIAL: NCT04739709
Title: A Multicenter, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of APP13007 for the Treatment of Inflammation and Pain After Cataract Surgery
Brief Title: Efficacy and Safety of APP13007 for Treatment of Inflammation and Pain After Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Formosa Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPN-301
Record Dates: First submitted 2021-01-26; First posted 2021-02-05 (Actual); Results first posted 2023-07-05 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Ocular Inflammation and Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APP13007 0.05% BID (Experimental): 1 drop APP13007 0.05% twice daily for 14 days to study (operated) eye
  Interventions: Drug: APP13007, 0.05%
- Matching Vehicle Placebo (Placebo Comparator): 1 drop matching vehicle place twice daily for 14 days to study (operated) eye
  Interventions: Drug: Matching Vehicle Placebo for APP13007, 0.05%

INTERVENTIONS:
Drug: APP13007, 0.05% — APP13007 eye drop, 0.05%
  Arms: APP13007 0.05% BID
Drug: Matching Vehicle Placebo for APP13007, 0.05% — Matching vehicle placebo eye drop
  Arms: Matching Vehicle Placebo

SUMMARY:
This Phase 3 study will evaluate APP13007 in comparison to the matching vehicle placebo in a randomized, parallel-group, double-masked fashion. The subjects will have undergone routine cataract surgery on Day 0 of the study and will be assessed the next day (Post-operative Day 1; POD1) after uncomplicated surgery for eligibility for randomization to study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older expected to undergo unilateral uncomplicated cataract extraction via phacoemulsification and posterior chamber intraocular lens implantation in one eye.
* Have a pin-hole corrected visual acuity without other correction of ≤ 1.3 logarithm of the minimum angle of resolution (logMAR) in the study eye to be operated and contralateral eye as measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart at Visit 1.
* Willing and able to comply with study requirements and visit schedule.
* Provide signed and dated informed consent.

Exclusion Criteria:

* Have a known sensitivity or allergy to clobetasol propionate, corticosteroids, or any of the study medication's components including benzalkonium chloride and soybean lecithin or any routine medication required during cataract surgery or for the conduct of study procedures
* Have an ACC count > 0 or any evidence of intraocular inflammation (e.g., flare) in either eye at the Screening visit
* Have a Grade > 0 on the Ocular Pain Assessment in either eye at the Screening visit

Note: Other inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (34):
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Global Research Management, Glendale, California
  - Inland Eye Specialists, Hemet, California
  - SoCal Eye Physicians and Associates, Long Beach, California
  - North Valley Eye Medical Group, Inc., Mission Hills, California
  - LoBue Laser and Eye Medical Center, Inc., Murrieta, California
  - Pendleton Eye Center, Oceanside, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Shasta Eye Medical Group, Inc., Redding, California
  - Icon Eye Care, Grand Junction, Colorado
  - Levenson Eye Associates, Jacksonville, Florida
  - International Eye Associates, PA, Ormond Beach, Florida
  - Newsom Eye and Laser Center, Sebring, Florida
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Jacksoneye SC, Columbus, Illinois
  - Midwest Cornea Associates, LLC, Carmel, Indiana
  - Senior Health Services, Louisville, Kentucky
  - Silverstein Eye Centers, PC, Kansas City, Missouri
  - Ophthalmology Consultants, Ltd., St Louis, Missouri
  - Comprehensive Eye Care, Ltd., Washington, Missouri
  - NV Eye Surgery, Henderson, Nevada
  - Center For Sight, Las Vegas, Nevada
  - Raymond Fong, MD, PC, New York, New York
  - Carolina Eye Associates, Southern Pines, North Carolina
  - Eye Physicians, LLC, Columbus, Ohio
  - Bucci Laser Vision Institute, Wilkes-Barre, Pennsylvania
  - Keystone Research Ltd., Austin, Texas
  - Retina Research Center, PLLC, Austin, Texas
  - Houston Eye Associates, Houston, Texas
  - Advanced Laser Vision and Surgical Institute, Houston, Texas
  - Lake Travis Eye and Laser Center, Lakeway, Texas
  - R and R Eye Research, LLC, San Antonio, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - Stacy R. Smith, MD, PC, Salt Lake City, Utah
- Centro Oftalmologico Metropolitano, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-center US study in which 27 sites recruited subjects between January 2021 and February 2022.
Pre-assignment Details: Of 456 enrolled participants, 378 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Started | 181 | 197
Completed | 180 | 197
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo | Total
Number analyzed (Participants) | 181 | 197 | 378
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (8.9) | 67.8 (8.6) | 68.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 119 | 225
  Male | 75 | 78 | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 52 | 87
  Not Hispanic or Latino | 146 | 145 | 291
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 11 | 16 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 27 | 45
  White | 150 | 151 | 301
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 181 | 197 | 378

OUTCOME MEASURES:

1. Primary Outcome: Participants With ACC Count = 0 at All Visits From Postoperative Day 8 Through Postoperative Day 15 Without Rescue Medication
Description: The number of cells in the anterior chamber of the eye are counted using slit-lamp biomicroscopy at each study visit and the results are reported as number of cells in a 1mm x 1mm area.
Time Frame: Postoperative Day 8 and Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
Participants | 48 | 10
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

2. Primary Outcome: Participants With Ocular Pain Grade = 0 at All Visits From Postoperative Day 4 Through Postoperative Day 15 Without Rescue Medication
Description: Ocular pain is measured in each eye using a subject-reported five-point (0-4) ocular pain grade scale (0 = no pain; 1 = minimal; 2 = mild; 3 = moderate; 4 = severe pain).
Time Frame: Postoperative Day 4, Postoperative Day 8 and Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
Participants | 123 | 46
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

3. Primary Outcome: Participants With Treatment-emergent Adverse Events (AEs)
Description: Number of participants with ocular and systemic treatment-emergent AEs.
Time Frame: From First dose to Postoperative Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
Participants | 38 | 39

4. Secondary Outcome: Participants With Anterior Chamber Cell Grade = 0 at POD8 Without Rescue Medication
Description: The number of cells in the anterior chamber of the eye are counted using slit-lamp biomicroscopy at each study visit and the results are reported as number of cells in a 1mm x 1mm area. ACC Grade 0 = 0 cells, ACC grade 1 = 1-5 cells, ACC grade 2 = 6-15 cells, ACC grade 3 = 16-30 cells, ACC grade 4 = >30 cells
Time Frame: Postoperative Day 8
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
Participants | 59 | 23
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

5. Secondary Outcome: Participants With Anterior Chamber Cell Grade = 0 at POD15 Without Rescue Medication
Description: as for outcome 4
Time Frame: Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
Participants | 106 | 31
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

6. Secondary Outcome: Participants With Ocular Pain Grade = 0 at POD4 Without Rescue Medication
Description: Ocular pain is measured in each eye using a subject-reported five-point (0-4) ocular pain grade scale (0 = no pain; 4 = severe pain).
Time Frame: Postoperative Day 4
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
Participants | 140 | 86
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

7. Secondary Outcome: Participants With Ocular Pain Grade = 0 at POD8 Without Rescue Medication
Description: as for outcome 6
Time Frame: Postoperative Day 8
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
Participants | 149 | 84
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

8. Secondary Outcome: Participants With Ocular Pain Grade = 0 at POD15 Without Rescue Medication
Description: as for outcome 6
Time Frame: Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
Participants | 164 | 83
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

9. Secondary Outcome: Participants With Anterior Chamber Flare (ACF) = 0 at POD4 Without Rescue Medication
Description: The degree of turbidity (flare) in the anterior chamber of the eye is measured using slit-lamp biomicroscopy and quantified on a five-point (0-4) anterior chamber flare grade scale (0 = none; 4 = Intense).
Time Frame: Postoperative Day 4
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
Participants | 111 | 79
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

10. Secondary Outcome: Participants With Anterior Chamber Flare (ACF) = 0 at POD8 Without Rescue Medication
Description: as for outcome 9
Time Frame: Postoperative Day 8
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
Participants | 142 | 75
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

11. Secondary Outcome: Participants With Anterior Chamber Flare (ACF) = 0 at POD15 Without Rescue Medication
Description: as for outcome 9
Time Frame: Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
Participants | 159 | 65
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

12. Secondary Outcome: Anterior Chamber Cell Grade - Change From Baseline (POD1 Prior to Dosing) to POD 15
Description: The number of cells in the anterior chamber of the eye are counted using slit-lamp biomicroscopy and the results are reported as number of cells in a 1mm x 1mm area using a 5 point grading scale. ACC Grade 0 = 0 cells, ACC grade 1 = 1-5 cells, ACC grade 2 = 6-15 cells, ACC grade 3 = 16-30 cells, ACC grade 4 = >30 cells
Time Frame: Baseline and Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: grade on a scale
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
grade on a scale | -2.1 (0.1) | -0.6 (0.1)
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -1.6, 95% CI 2-sided [-1.8 to -1.3] — Treatment Difference = APP13007-Placebo. Mean Difference Is the least-squares mean difference from the ANCOVA model with treatment as a fixed effect and baseline as a covariate

13. Secondary Outcome: Ocular Pain Grade - Change From Baseline (POD1 Prior to Dosing) to POD 15
Description: as for outcome 6
Time Frame: Baseline and Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: grade on a scale
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
grade on a scale | -1.1 (0.1) | -0.3 (0.1)
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-0.9 to -0.6] — [estimate comment as in outcome 12, analysis 1]

14. Secondary Outcome: Anterior Chamber Flare (ACF) - Change From Baseline (POD1 Prior to Dosing) to POD 15
Description: as for outcome 9
Time Frame: Baseline and Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: grade on a scale
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
grade on a scale | -0.7 (0.1) | -0.0 (0.0)
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-0.8 to -0.5] — [estimate comment as in outcome 12, analysis 1]

15. Secondary Outcome: Best Corrected Visual Acuity - Change From Baseline (POD1 Prior to Dosing) to POD4
Description: The visual acuity in each eye is corrected using the pinhole method and the acuity is quantified on a logMAR (minimal angle of resolution) scale using the 'Early Treatment Diabetic Retinopathy Study' [ETDRS] charts for right and left eyes.
  A logMAR Score is calculated using the letter row on the chart and the number of incorrect letters read by the participant.
Time Frame: Baseline and Postoperative Day 4
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: logMAR score
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
logMAR score | -0.07 (0.01) | -0.04 (0.01)
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p = 0.017, ANCOVA; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.06 to -0.01] — [estimate comment as in outcome 12, analysis 1]

16. Secondary Outcome: Best Corrected Visual Acuity - Change From Baseline (POD1 Prior to Dosing) to POD8
Description: as for outcome 15
Time Frame: Baseline and Postoperative Day 8
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: logMAR score
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
logMAR score | -0.10 (0.01) | -0.02 (0.01)
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.10 to -0.04] — [estimate comment as in outcome 12, analysis 1]

17. Secondary Outcome: Best Corrected Visual Acuity - Change From Baseline (POD1 Prior to Dosing) to POD15
Description: as for outcome 15
Time Frame: Baseline and Postoperative Day 15
Population: Intent to Treat Population. Last observation carried forward (LOCF) imputation method.
Measure: Least Squares Mean (Standard Error); unit: logMAR score
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
logMAR score | -0.11 (0.01) | -0.02 (0.01)
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.11 to -0.06] — [estimate comment as in outcome 12, analysis 1]

18. Secondary Outcome: Participants Using of Anti-inflammatory 'Rescue' Medication Through End-of-Treatment
Description: Participants who do not respond to study treatment after randomization are started on anti-inflammatory medication (referred to as 'Rescue' medication). The number of subjects starting 'Rescue' medication is recorded at each study visit
Time Frame: First dose to Postoperative Day 15
Population: Intent to Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
Number analyzed (Participants) | 181 | 197
Participants | 10 | 100
Statistical Analysis 1: Comparison: APP13007 0.05% BID vs Matching Vehicle Placebo; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: All-Cause Mortality data were collected from informed consent through Postoperative Day 22. Serious adverse events were collected from informed consent through Postoperative Day 22. Other (not Including Serious) adverse events were collected from the first dose through Postoperative Day 22.
Arm/Group | APP13007 0.05% BID | Matching Vehicle Placebo
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/197
Serious Adverse Events (participants affected / at risk) | 0/181 | 0/197
Other Adverse Events (participants affected / at risk) | 3/181 | 10/197
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APP13007 0.05% BID (N=181) | Matching Vehicle Placebo (N=197)
Corneal oedema (Eye disorders) | 3 (3) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institutions and Investigators participating in this trial shall have no right to publish or present the results of this study without the prior written consent of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/09/NCT04739709/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04739709/SAP_001.pdf